CLINICAL TRIAL: NCT03910023
Title: Non-pharmacological Treatment for Chronic Back Pain: a Randomised, Controlled Trial
Brief Title: Non-pharmacological Treatment for Chronic Back Pain
Acronym: LOMBATHERM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-A02801-54
Record Dates: First submitted 2019-03-12; First posted 2019-04-10 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-06

CONDITIONS: Low Back Pain
Keywords: Low back pain; Crenobalneotherapy; Spa therapy; Mud application; Water exercises; Underwater massages
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: In this prospective, evaluator-blinded, multi-centre, 2-parallel-arm, Zelen randomized (1:1), controlled trial, UCHE alone will be compared to spa therapy in addition to UCHE for the treatment of chronic low back pain.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group will perform home exercises alone
  Interventions: Other: Usual care comporting a home-exercise program (UCHE)
- Spa group (Experimental): The spa group will be proposed an additional spa treatment
  Interventions: Other: Usual care comporting a home-exercise program (UCHE); Other: Spa therapy

INTERVENTIONS:
Other: Usual care comporting a home-exercise program (UCHE) — The UCHE intervention will correspond to current practice (including the continuation of previous treatments, if applicable) as decided by the attending physician. The patient will also be provided with a practical guide on how to manage back pain (the "back book"), including a recommended home exercise program.
Other: Spa therapy — the spa-therapy intervention consists of 18 consecutive days of spa-therapy (excepting Sundays), that must occur with 60 days of randomisation. The latter will combine mineral water with physical and hydrotherapeutic treatments, including massages, heat and water exercises.
  Arms: Spa group

SUMMARY:
The working hypothesis is that spa therapy in addition to usual care including home exercises (UCHE) will result in greater improvements in pain reduction, associated disability and quality of life for chronic low back pain patients. It follows that health resource consumption and linked costs should also be reduced. The primary objective of this study is therefore to compare the therapeutic effect of UCHE alone versus spa therapy in addition to UCHE for chronic low back pain.

DETAILED DESCRIPTION:
Secondarily, the study will also (i) evaluate the therapeutic effects specific to each spa-centre, (ii) specifically describe effects among subjects who are currently engaged in a professional activity, (iii) evaluate treatment tolerance as well as (iv) per-patient health resource use and associated costs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient presenting with chronic low back pain: usual pain of the lumbar region lasting for more than 3 months. This pain may radiate to the buttocks, iliac crest, and does not go past the knee.
* Patient presenting with a current pain intensity on a visual analogue scale (VAS) > or = 40 mm.
* The patient has signed the informed consent
* The patient is a beneficiary of a social security programme [national health insurance]

Exclusion Criteria:

* Patients with secondary low back pain
* Patients with severe depression, psychosis
* Patients who have already had a spa treatment in the previous 6 months
* Patients with a contraindication for spa treatment
* Patients with a professional activity related to hydrotherapy (to avoid any conflict of interest)
* Patients with sciatic pain beyond the knee (sciatica being a non-indication for spa treatment)
* Other treatments that may interact according to the judgment of the investigator
* Patients who live more than 30 km away from the spa

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Presence/absence of a clinically relevant change in visual analogue scale (VAS) score for pain | 6 months
  Presence/absence of a clinically relevant change in visual analogue scale (VAS) score for pain, defined by an improvement of at least 30%; cases where patients demonstrate a 30% improvement in VAS scores for pain but nevertheless require hospitalisation for back pain during the study follow-up period will be considered as treatment failures (absence of clinically relevant change).

SECONDARY OUTCOMES:
Huskinsson's VAS for pain. | Baseline (day 0)
Huskinsson's VAS for pain. | 1 month
Huskinsson's VAS for pain. | 6 months
Huskinsson's VAS for pain. | 12 months
The EIFEL scale | Baseline (day 0)
  The EIFEL scale: the validated French version of a disability rating scale by Rolland and Morris. This 24-question scale (with scores ranging from 0 (no impact) to 24 (maximum impact) quantifies the impact of low back pain on daily life.
The EIFEL scale | 1 month
  The EIFEL scale: the validated French version of a disability rating scale by Rolland and Morris. This 24-question scale (with scores ranging from 0 (no impact) to 24 (maximum impact) quantifies the impact of low back pain on daily life.
The EIFEL scale | 6 months
  The EIFEL scale: the validated French version of a disability rating scale by Rolland and Morris. This 24-question scale (with scores ranging from 0 (no impact) to 24 (maximum impact) quantifies the impact of low back pain on daily life.
The EIFEL scale | 12 months
  The EIFEL scale: the validated French version of a disability rating scale by Rolland and Morris. This 24-question scale (with scores ranging from 0 (no impact) to 24 (maximum impact) quantifies the impact of low back pain on daily life.
The Fear Avoidance and Belief Questionnaire (FABQ) | Baseline (day 0)
  The Fear Avoidance and Belief Questionnaire (FABQ) assess inappropriate fears and beliefs concerning back pain; the validated French version will be used.
The Fear Avoidance and Belief Questionnaire (FABQ) | 1 month
  The Fear Avoidance and Belief Questionnaire (FABQ) assess inappropriate fears and beliefs concerning back pain; the validated French version will be used.
The Fear Avoidance and Belief Questionnaire (FABQ) | 6 months
  The Fear Avoidance and Belief Questionnaire (FABQ) assess inappropriate fears and beliefs concerning back pain; the validated French version will be used.
The Fear Avoidance and Belief Questionnaire (FABQ) | 12 months
  The Fear Avoidance and Belief Questionnaire (FABQ) assess inappropriate fears and beliefs concerning back pain; the validated French version will be used.
The EQ-5D-5L questionnaire | Baseline (day 0)
  The EQ-5D-5L questionnaire will be used to track changes in quality of life. This self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
The EQ-5D-5L questionnaire | 1 month
  The EQ-5D-5L questionnaire will be used to track changes in quality of life. This self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
The EQ-5D-5L questionnaire | 6 months
  The EQ-5D-5L questionnaire will be used to track changes in quality of life. This self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
The EQ-5D-5L questionnaire | 12 months
  The EQ-5D-5L questionnaire will be used to track changes in quality of life. This self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Patient Acceptable Symptom State (PASS) | Baseline (day 0)
  Patient Acceptable Symptom State (PASS): Yes/no response to the following question: "If you take into account all the activities you have in your daily life, the importance of your pain and your disability, do you consider your condition as satisfactory?"
Patient Acceptable Symptom State (PASS) | 1 month
  Patient Acceptable Symptom State (PASS): Yes/no response to the following question: "If you take into account all the activities you have in your daily life, the importance of your pain and your disability, do you consider your condition as satisfactory?"
Patient Acceptable Symptom State (PASS) | 6 months
  Patient Acceptable Symptom State (PASS): Yes/no response to the following question: "If you take into account all the activities you have in your daily life, the importance of your pain and your disability, do you consider your condition as satisfactory?"
Patient Acceptable Symptom State (PASS) | 12 months
  Patient Acceptable Symptom State (PASS): Yes/no response to the following question: "If you take into account all the activities you have in your daily life, the importance of your pain and your disability, do you consider your condition as satisfactory?"
Overall opinion of the patient on his/her state of health (5-point Likert scale) | Baseline (day 0)
  Overall opinion of the patient on his/her state of health (5-point Likert scale)
Overall opinion of the patient on his/her state of health (5-point Likert scale) | 1 month
  Overall opinion of the patient on his/her state of health (5-point Likert scale)
Overall opinion of the patient on his/her state of health (5-point Likert scale) | 6 months
  Overall opinion of the patient on his/her state of health (5-point Likert scale)
Overall opinion of the patient on his/her state of health (5-point Likert scale) | 12 months
  Overall opinion of the patient on his/her state of health (5-point Likert scale)
Overall opinion of the evaluating physician on the patient's state of health (5-point Likert scale) | Baseline (day 0)
  Overall opinion of the evaluating physician on the patient's state of health (5-point Likert scale)
Overall opinion of the evaluating physician on the patient's state of health (5-point Likert scale) | 1 month
  Overall opinion of the evaluating physician on the patient's state of health (5-point Likert scale)
Overall opinion of the evaluating physician on the patient's state of health (5-point Likert scale) | 6 months
  Overall opinion of the evaluating physician on the patient's state of health (5-point Likert scale)
Overall opinion of the evaluating physician on the patient's state of health (5-point Likert scale) | 12 months
  Overall opinion of the evaluating physician on the patient's state of health (5-point Likert scale)
Daily drug consumption over the past 72 hours: Analgesics | Baseline (day 0)
  Daily drug consumption over the past 72 hours: Analgesics (in mg of paracetamol and morphine equivalents).
Daily drug consumption over the past 72 hours: Analgesics | 1 month
  Daily drug consumption over the past 72 hours: Analgesics (in mg of paracetamol and morphine equivalents).
Daily drug consumption over the past 72 hours: Analgesics | 6 months
  Daily drug consumption over the past 72 hours: Analgesics (in mg of paracetamol and morphine equivalents).
Daily drug consumption over the past 72 hours: Analgesics | 12 months
  Daily drug consumption over the past 72 hours: Analgesics (in mg of paracetamol and morphine equivalents).
Daily drug consumption over the past 72 hours: NSAIDs | Baseline (day 0)
  Daily drug consumption over the past 72 hours: NSAIDs (reported in mg and as a percentage of the maximum dose)
Daily drug consumption over the past 72 hours: NSAIDs | 1 month
  Daily drug consumption over the past 72 hours: NSAIDs (reported in mg and as a percentage of the maximum dose)
Daily drug consumption over the past 72 hours: NSAIDs | 6 months
  Daily drug consumption over the past 72 hours: NSAIDs (reported in mg and as a percentage of the maximum dose)
Daily drug consumption over the past 72 hours: NSAIDs | 12 months
  Daily drug consumption over the past 72 hours: NSAIDs (reported in mg and as a percentage of the maximum dose)
Daily drug consumption over the past 72 hours: Corticosteroids | Baseline (day 0)
  Daily drug consumption over the past 72 hours: Corticosteroids (in mg equivalent prednisone)
Daily drug consumption over the past 72 hours: Corticosteroids | 1 month
  Daily drug consumption over the past 72 hours: Corticosteroids (in mg equivalent prednisone)
Daily drug consumption over the past 72 hours: Corticosteroids | 6 months
  Daily drug consumption over the past 72 hours: Corticosteroids (in mg equivalent prednisone)
Daily drug consumption over the past 72 hours: Corticosteroids | 12 months
  Daily drug consumption over the past 72 hours: Corticosteroids (in mg equivalent prednisone)
Daily drug consumption over the past 72 hours: Benzodiazepine muscle relaxants: | Baseline (day 0)
  Daily drug consumption over the past 72 hours: Benzodiazepine muscle relaxants: % of maximum dose
Daily drug consumption over the past 72 hours: Benzodiazepine muscle relaxants: | 1 month
  Daily drug consumption over the past 72 hours: Benzodiazepine muscle relaxants: % of maximum dose
Daily drug consumption over the past 72 hours: Benzodiazepine muscle relaxants: | 6 months
  Daily drug consumption over the past 72 hours: Benzodiazepine muscle relaxants: % of maximum dose
Daily drug consumption over the past 72 hours: Benzodiazepine muscle relaxants: | 12 months
  Daily drug consumption over the past 72 hours: Benzodiazepine muscle relaxants: % of maximum dose
Number of infiltrations | 12 months
Estimated per-patient cost for one year of care | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche rhumatologique et thermal, Aix-les-Bains, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to, in as much as possible, make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  Due to conditions imposed by French law, data will be made available to the public upon request to the AFRETH scientific committee (Association Française pour la Recherche Thermale, 1 rue Cels 75014 Paris, France; http://www.afreth.org).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: As close to "real time" as possible, the following supporting information will be made public:
  * Study Protocol
  * Statistical Analysis Plan
  * Participant Information materials
  * Analytic code
  The study protocol will be submitted to the journal "Trials" for publication.
  The remaining documents will either be published or posted / registered on osf.io/clinicaltrials.gov. The clinicaltrials.gov registration will contain a link that points to the appropriate osf.io page.
  Requests for individual datasets can be made anytime following full publication of results.
Access Criteria: Due to French law there are restrictions on publicly sharing the data of this study. Data requests may be submitted to the AFRETH and must be approved by the French data protection authority, la Commission Nationale de l'Informatique et des Libertés. Data requests may be sent to AFRETH. French law requires that everyone who wishes to access cohorts data or clinical study data on humans must ask the French data protection authority, la Commission Nationale de l'Informatique et des Libertés (CNIL), for permission. For further information, please see: https://www.cnil.fr/. "
URL: https://osf.io/ahpwy/

REFERENCES:
- [Derived] Forestier R, Suehs C, Francon A, Marty M, Genevay S, Sellam J, Chauveton C, Erol Forestier FB, Molinari N. Usual care including home exercise with versus without spa therapy for chronic low back pain: protocol for the LOMBATHERM' study, a multicentric randomised controlled trial. Trials. 2020 May 11;21(1):392. doi: 10.1186/s13063-020-04271-9. PMID 32393320